CLINICAL TRIAL: NCT05043545
Title: Evaluation and Application of Experimental Indices for the Study of Potential Prognostic Factors in Patients With Acute Neurological Injury, Using Low-frequency Sampled Data
Brief Title: Long Pressure Autoregulation Index
Acronym: Long PAx
Status: Completed | Type: Observational
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Paolo GRITTI, Principal Investigator, Papa Giovanni XXIII Hospital
Other Study IDs: PapaGiovanni H
Record Dates: First submitted 2021-08-29; First posted 2021-09-14 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pressure reactivity index (PRx) has emerged as a surrogate method for the continuous bedside estimation of global cerebral autoregulation and a significant predictor of unfavorable outcomes. However, calculations require continuous, high-resolution monitoring and are currently limited to specialized ICUs with dedicated software. To overcome this problem, new indices calculated using one-minute average data, instead of 10-second average data as performed by the PRx, have been proposed.

The study aims to test new physiological indices appropriately modified to adapt to the scarcity of output data generated by standard hospital systems (frequency ~0.0033 Hz, approximately a 5-minute period) and to evaluate their association with outcome measures.

DETAILED DESCRIPTION:
Data preparation and index calculations were performed using an in-house algorithm.

Data extracted and processed with the algorithm:

Ultra-low pressure reactivity index (UL-PRx), Intracranial pressure (ICP), Cerebral perfusion pressure (CPP), Arterial blood pressure (ABP), heart rate (HR), respiratory rate (RR), temperature, end-tidal CO2 (EtCO2), saturation (SpO2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of acute neurological injury requiring intracranial pressure (ICP) monitoring.
* Availability of continuous intensive care monitoring of physiological data.

Exclusion Criteria:

Patients with less than 8 hours of physiological data monitoring.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute neurological injury admitted to ICU of the ASST Papa Giovanni XXIII requiring ICP monitoring during the study period (January 2013 - June 2022). For Traumatic Brain Injury (TBI) it is estimated that medical records from approximately 210 TBI subjects requiring ICP monitoring will be reviewed. The final number of subjects to be included will be determined based on available medical records obtained within the timeframe of the estimated duration of the study.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
mortality | 12-months
  The binary outcome of mortality (dead vs alive) during hospitalization and at 12-months
Glasgow Outcome Scale - Extended (GOSE) | 12-months
  The global functional outcome at 12 months assessed by Glasgow Outcome Scale-Extended (GOS-E), dichotomized into favorable (a score of 5-6 defines a score of 5 to 8, Moderate Disability) and unfavorable (a score of 1 to 4, Dead is characterized by a score of 1).

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Gritti, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gritti P, Bonfanti M, Zangari R, Bonanomi E, Di Matteo M, Dell'Avanzo G, Corbella D, Micheli F, Lanterna LA, Lando G, Pezzetti G, Vascello MF, Biroli F, Lorini FL. Visualizing and Interpreting the Carbon Dioxide Reactivity Index in Traumatic Brain Injury. Neurocrit Care. 2026 Jan 8. doi: 10.1007/s12028-025-02429-4. Online ahead of print. PMID 41507673
- [Derived] Gritti P, Bonfanti M, Zangari R, Bonanomi E, Di Matteo M, Corbella D, Farina A, Lecchi L, Togni T, Mandelli P, Lanterna LA, Biroli F, Lorini FL. Continuous monitoring of intracranial pressure and end tidal carbon dioxide variations in traumatic brain injury: introducing the carbon dioxide reactivity index (CO2Rx). J Clin Monit Comput. 2025 Jun;39(3):581-594. doi: 10.1007/s10877-025-01285-z. Epub 2025 Mar 22. PMID 40120011
- [Derived] Gritti P, Bonfanti M, Zangari R, Bonanomi E, Farina A, Pezzetti G, Pelliccioli I, Longhi L, Di Matteo M, Viscone A, Lando G, Cavalleri G, Gerevini S, Biroli F, Lorini FL. Cerebral autoregulation in traumatic brain injury: ultra-low-frequency pressure reactivity index and intracranial pressure across age groups. Crit Care. 2024 Jan 23;28(1):33. doi: 10.1186/s13054-024-04814-5. PMID 38263241
- [Derived] Gritti P, Bonfanti M, Zangari R, Bonanomi E, Pellicioli I, Mandelli P, Longhi L, Rasulo FA, Bertuetti R, Farina A, Biroli F, Lorini FL. Evaluation and application of ultra-low-frequency pressure reactivity index in pediatric traumatic brain injury patients. Acta Neurochir (Wien). 2023 Apr;165(4):865-874. doi: 10.1007/s00701-023-05538-1. Epub 2023 Feb 27. PMID 36847979